CLINICAL TRIAL: NCT07314983
Title: Report of a Clinical-biological Case: "Long-term Anticoagulation in a Patient With Severe Hemophilia A
Brief Title: Long-term Anticoagulation in a Patient With Severe Hemophilia A
Acronym: HAAC
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9816
Record Dates: First submitted 2025-09-22; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-09

CONDITIONS: Hemophilia A
Keywords: Hemophilia A; Severe Hemophilia A; factor VIII (FVIII) deficiency; Antithrombotic protection; Anticoagulant therapy
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To date, and to our knowledge, no case of severe hemophilia A patients receiving long-term anticoagulation has been published. Severe hemophilia A is a hereditary bleeding disorder characterized by a factor VIII (FVIII) deficiency of <1%. Anticoagulation remains a real challenge in these patients, given the precarious hemostatic balance between the bleeding risk associated with anticoagulation and the antithrombotic protection associated with factor VIII deficiency. The advent of new replacement therapies, characterized by FVIII molecules with a prolonged or very prolonged half-life, provides a high level of FVIII coverage (and therefore protection against the risk of bleeding) in patients receiving prophylaxis, thus facilitating the initiation of anticoagulation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years) with severe hemophilia A
* Absence of written objection in the subject's medical record to the reuse of their data for scientific research purposes.

Exclusion Criteria:

- Subject having expressed objection to the reuse of their data for scientific research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient (≥ 18 years) with severe hemophilia A
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
FVIII Level | Up to 15 months
  Factor VIII (FVIII) is a clotting protein: it enables the blood to form a clot to stop bleeding.
  Its level indicates how well the blood clots, which is useful for diagnosing or monitoring hemophilia A before surgery.
  General values:
  * Normal: approximately 50 to 150%
  * Too low: risk of bleeding
  * Too high: may increase the risk of clots

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratoire d'Hématologie - Unité d'Hémostase - CHU de Strasbourg - France, Strasbourg, France